CLINICAL TRIAL: NCT05475002
Title: A Randomized Controlled Trial of a Care Empowerment Program Using Virtual Reality for Family Caregivers of People With Dementia
Brief Title: A Care Empowerment Program Using Virtual Reality for Family Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Huei-Chuan Sung, Associate professor, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YLH-IRB-11104
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Dementia Family Caregiver
Keywords: family caregiver; dementia; virtual reality; empowerment
MeSH Terms: conditions — Dementia; Empowerment

STUDY DESIGN:
Intervention Model Description: two-group randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): care empowerment program
  Interventions: Other: care empowerment program
- Control group (Active Comparator): routine family support
  Interventions: Other: Routine family support

INTERVENTIONS:
Other: care empowerment program — dementia care e-books and dementia virtual reality activity in addition to the routine dementia care manual and family support group
  Arms: Intervention group
Other: Routine family support — routine dementia care manual and family support group
  Arms: Control group

SUMMARY:
This study aims to evaluate a care empowerment program using virtual reality on dementia knowledge, attitude, self-efficacy in managing BPSD, empathy and caregiver burden of family caregivers of people with dementia.

DETAILED DESCRIPTION:
The majority of patients with dementia live at home and cared by their families in Taiwan. Most of family caregivers have limited knowledge and care skills of dementia, therefore they experience great stress and caregiver burden which may have negative impact on their physical and mental health.

This two-group randomised controlled trial aims to evaluate a care empowerment program using virtual reality on dementia knowledge, attitude, care self-efficacy in managing BPSD, empathy and caregiver burden of family caregivers of people with dementia.

The intervention group will receive the Care Empowerment Program, which consists of dementia care e-books and virtual reality-based dementia activities, in addition to the routine dementia care manual and family support group.

The control group will only receive routine dementia care manual and family support group with no dementia virtual reality activity.

Both groups will be assessed for their dementia knowledge, attitudes, self-efficacy in managing BPSD, empathy and caregiver burden at baseline, month 3, and 4.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 90 years,
* Taiwanese nationality,
* have provided care for relatives with dementia or cognitive impairment for at least three months,
* have a mobile phone or tablet and regular access to the internet,
* provide informed consent to participate in the study.

Exclusion Criteria:

* family members who do not meet the inclusion criteria,
* can not provide informed consent.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale (DKAS) | baseline
  score of knowledge about dementia
Dementia Knowledge Assessment Scale (DKAS) | month 3
  score of knowledge about dementia
Dementia Knowledge Assessment Scale (DKAS) | month 4
  score of knowledge about dementia
Approaches to Dementia Questionnaire (ADQ) | baseline
  score of attitude toward people with dementia
Approaches to Dementia Questionnaire (ADQ) | month 3
  score of attitude toward people with dementia
Approaches to Dementia Questionnaire (ADQ) | month 4
  score of attitude toward people with dementia
Family Caregiver Competence Questionnaire (FACCQ) | baseline
  score of FACCQ
Family Caregiver Competence Questionnaire (FACCQ) | month 3
  score of FACCQ
Family Caregiver Competence Questionnaire (FACCQ) | month 4
  score of FACCQ
Revised Interpersonal Reactivity Index (R-IRI) | baseline
  empathy toward people with dementia
Revised Interpersonal Reactivity Index (R-IRI) | month 3
  empathy toward people with dementia
Revised Interpersonal Reactivity Index (R-IRI) | month 4
  empathy toward people with dementia

SECONDARY OUTCOMES:
Caregiver Burden Inventory (CBI) | baseline
  score of caregiver burden for caring for people with dementia
Caregiver Burden Inventory (CBI) | month 3
  score of caregiver burden for caring for people with dementia
Caregiver Burden Inventory (CBI) | month 4
  score of caregiver burden for caring for people with dementia

CONTACTS AND LOCATIONS:
Locations (1):
- TCU dementia day center, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No